CLINICAL TRIAL: NCT04669665
Title: A 2-part Phase 2 Study to Assess the Efficacy, Safety, and Tolerability of SLS-002 (Intranasal Racemic Ketamine) Administered to Adults With Major Depressive Disorder at Imminent Risk of Suicide
Brief Title: A Study of SLS-002 (Intranasal Racemic Ketamine) in Adults With Major Depressive Disorder at Imminent Risk of Suicide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seelos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLS-002-201
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Depressive Disorder, Major; Suicidal
Keywords: Depression; Depressive disorder; SLS-002; Mental disorders; Suicide; Suicidal Ideation; Mood disorders; Behavioral symptoms; Self-injurious behavior; Ketamine; Antidepressive agents; Psychotropic drugs
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder; Mental Disorders; Suicide; Suicidal Ideation; Mood Disorders; Behavioral Symptoms; Self-Injurious Behavior | interventions — Ketamine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Part 1 is a single group. Part 2 is a parallel group 1:1 randomization of SLS-002 to placebo, plus standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 is open-label. Part 2 is a double-blind placebo-controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SLS-002 + Standard of care (Experimental): Participants will receive SLS-002 (intranasal racemic ketamine) 90 milligram (mg) two times per week for 2 weeks with standard of care treatment
  Interventions: Drug: SLS-002; Other: Standard of care; Device: Intranasal device
- Placebo + Standard of care (Placebo Comparator): Participants will receive intranasal placebo two times per week for 2 weeks with standard of care treatment
  Interventions: Drug: Placebo; Other: Standard of care; Device: Intranasal device

INTERVENTIONS:
Drug: SLS-002 — Intranasal racemic ketamine hydrochloride 90 milligrams (mg)
  Other Names: Ketamine hydrochloride
  Arms: SLS-002 + Standard of care
Drug: Placebo — Intranasal placebo
  Arms: Placebo + Standard of care
Other: Standard of care — Standard of care treatment will be determined by the treating physician(s) based on clinical judgement and practice guidelines
Device: Intranasal device — Device to deliver intranasal solution

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, and tolerability of SLS-002 (intranasal racemic ketamine) in addition to standard of care on symptoms of Major Depressive Disorder (MDD) and suicidality, in participants who are assessed to be at imminent risk for suicide, as measured by the change from baseline on the Montgomery-Asberg Depression Rating Scale (MADRS) total score at 24 hours post first dose.

DETAILED DESCRIPTION:
This is a 2-part study: Part 1 is open-label, while Part 2 is a randomized, double-blind, placebo-controlled, multicenter study. The study will enroll participants with MDD for whom a physician has assessed to be at risk for suicide. The study will consist of a screening evaluation, a treatment period, and a safety follow-up period. Participants' safety will be evaluated throughout the study. If you or a loved one are having thoughts of suicide, please seek immediate medical help. Go to the emergency room or call the National Suicide Prevention Lifeline at 1-800-273-8255.

Potential participants may visit http://frontiersstudy.com/

ELIGIBILITY:
Inclusion Criteria:

* Participant with diagnosis of current MDD (unipolar without psychotic features) per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), with symptoms present for at least 4 weeks, based on psychiatric intake and confirmed by the Mini International Psychiatric Interview Version 7.02 for Suicidality Disorders (MINI).
* Participant has a Montgomery Åsberg Depression Rating Scale (MADRS) total score of ≥28 predose on Day 1, and has a score of 5 or 6 on item 10.
* Participant has a Clinical Global Impression of Severity for Suicidal Ideation and Behavior (CGIS-SI/B) score of ≥4 predose on Day 1.
* Participant requires psychiatric hospitalization due to significant risk of suicide, has ≥15 on the S-STS CMCM total score, and a score of 6-9 (inclusive) on the S-STS CMCM Clinician judgment of subject's risk of a suicide attempt or death by suicide at this time.
* Participant has a history of previous suicide attempt(s), as confirmed on the Columbia Suicide Severity Rating Scale (C-SSRS) with a history of at least one actual attempt, or if the attempt was interrupted or aborted, is judged to have been serious in intent.
* Participant is willing and able to take prescribed non-investigational antidepressant therapy(ies) at investigator's discretion for at least the duration of the study.

Exclusion Criteria:

* Participant has seizures, intellectual disability, a neurocognitive disorder or a lifetime diagnosis of bipolar disorder, any mood disorder with psychotic features, schizophrenia or other psychotic disorder, obsessive compulsive disorder, or antisocial personality disorder.
* In the investigator's opinion, participant has chronic, refractory treatment-resistant depression from >4 adequate therapeutic trials of antidepressants (with or without adjuvants and/or ECT) as confirmed by Antidepressant Treatment Response Questionnaire (ATRQ).
* Participant has a body mass index (BMI) >40 or <18 at screening, uncontrolled hypertension, or any clinically significant medical condition that might confound the results.
* Participant meets the DSM-5 criteria for moderate or severe substance use disorder or a positive urine test for drugs of abuse.
* Participant does not meet or is not willing to comply with the requirements listed in prohibited and restricted medications and therapies in the protocol, as well as required washout periods prior to participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at 24 Hours Post First Dose | Baseline (Day 1, predose) and 24 hours post first dose (Day 2)
  MADRS is clinician-rated scale designed to be used in participants with Major Depressive Disorder (MDD) to measure depression severity and detect changes due to antidepressant treatment. It evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic and suicidal thoughts. Scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms), summed for total possible score of 0 to 60.

SECONDARY OUTCOMES:
Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Day 16 | Baseline (Day 1, predose) and 2 weeks post first dose (Day 16)
  MADRS is clinician-rated scale designed to be used in participants with Major Depressive Disorder (MDD) to measure depression severity and detect changes due to antidepressant treatment. It evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic and suicidal thoughts. Scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of symptoms), summed for total possible score of 0 to 60.
Change From Baseline in Clinical Global Impression of Severity for Suicidal Ideation and Behavior (CGIS-SI/B) Scale at 24 Hours Post First Dose | Baseline (Day 1, predose) and 24 hours post first dose (Day 2)
  Clinical global impression of severity for suicidal ideation and behavior (CGIS-SI/B) scale is revised version of the clinical global impression severity scale (CGI-S), a global rating scale that gives an overall measure of the severity of a participant's illness. The CGIS-SI/B summarizes the clinician's overall impression of severity of suicidal ideation and behavior on a 5-point scale from 1 (not at all suicidal) to 5 (among the most extremely suicidal), based on the totality of information available to the clinician.
Change From Baseline in Patient Global Impression of Severity for Suicidal Ideation and Behavior (PGIS-SI/B) Scale at 24 Hours Post First Dose | Baseline (Day 1, predose) and 24 hours post first dose (Day 2)
  Patient global impression of severity for suicidal ideation and behavior (PGIS-SI/B) scale is revised version of the patient global impression severity scale (PGI-S), a global rating scale that gives the patient's perspective on their overall severity of suicidal impulses, thoughts, and behaviors. The PGIS-SI/B summarizes the patient's overall impression of severity of suicidal ideation and behavior on a 5-point scale from 1 (not present) to 5 (extremely severe).
Change From Baseline in Clinical Global Impression of Severity for Suicidal Ideation and Behavior (CGIS-SI/B) Scale at Day 16 | Baseline (Day 1, predose) and 2 weeks post first dose (Day 16)
  Clinical global impression of severity for suicidal ideation and behavior (CGIS-SI/B) scale is revised version of the clinical global impression severity scale (CGI-S), a global rating scale that gives an overall measure of the severity of a participant's illness. The CGIS-SI/B summarizes the clinician's overall impression of severity of suicidal ideation and behavior on a 5-point scale from 1 (not at all suicidal) to 5 (among the most extremely suicidal), based on the totality of information available to the clinician.
Change from Baseline in Sheehan-Suicidality Tracking Scale Clinically Meaningful Change Measure (S-STS CMCM) Total Score at 24 hours post first dose (Day 2) | Baseline (Day 1, predose) and 24 hours post first dose (Day 2)
  The Sheehan-Suicidality Tracking Scale Clinically Meaningful Change Measure (S-STS CMCM) is a clinician-rated outcome measure which assesses suicidal ideation and behavior on a standard 22-item scale, as well as multiple patient and clinician-rated items. The first 16 items are rated on a Likert-type scale ranging from 0 = not at all to 4 = extremely, where select scoring (i.e., 4 specific items are scored based on the highest score on 2 of those items) yields a total score ranging from 0 to 52.
Change From Baseline in Patient Global Impression of Severity for Suicidal Ideation and Behavior (PGIS-SI/B) Scale at Day 16 | Baseline (Day 1, predose) and 2 weeks post first dose (Day 16)
  Patient global impression of severity for suicidal ideation and behavior (PGIS-SI/B) scale is revised version of the patient global impression severity scale (PGI-S), a global rating scale that gives the patient's perspective on their overall severity of suicidal impulses, thoughts, and behaviors. The PGIS-SI/B summarizes the patient's overall impression of severity of suicidal ideation and behavior on a 5-point scale from 1 (not present) to 5 (extremely severe).
Change from Baseline in Sheehan-Suicidality Tracking Scale Clinically Meaningful Change Measure (S-STS CMCM) Total Score at Day 16 | Baseline (Day 1, predose) and 2 weeks post first dose (Day 16)
  The Sheehan-Suicidality Tracking Scale Clinically Meaningful Change Measure (S-STS CMCM) is a clinician-rated outcome measure which assesses suicidal ideation and behavior on a standard 22-item scale, as well as multiple patient and clinician-rated items. The first 16 items are rated on a Likert-type scale ranging from 0 = not at all to 4 = extremely.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Seelos Investigational Site, Orange, California
  - Seelos Investigational Site, Panorama City, California
  - Seelos Investigational Site, San Diego, California
  - Seelos Investigational Site, Hollywood, Florida
  - Seelos Investigational Site, Miami, Florida
  - Seelos Investigational Site, Miami Lakes, Florida
  - Seelos Investigational Site, Miramar, Florida
  - Seelos Investigational Site, Oakland Park, Florida
  - Seelos Investigational Site, Atlanta, Georgia
  - Seelos Investigational Site, Decatur, Georgia
  - Seelos Investigational Site, Springfield, Illinois
  - Seelos Investigational Site, Gaithersburg, Maryland
  - Seelos Investigational Site, Flowood, Mississippi
  - Seelos Investigational Site, Buffalo, New York
  - Seelos Investigational Site, Cincinnati, Ohio
  - Seelos Investigational Site, North Canton, Ohio
  - Seelos Investigational Site, DeSoto, Texas
  - Seelos Investigational Site, Houston, Texas
  - Seelos Investigational Site, Richardson, Texas
  - Seelos Investigational Site, Salt Lake City, Utah
  - Seelos Investigational Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.